# **©** RUSH

# CONSENT/AUTHORIZATION FOR PARTICIPATION IN A RESEARCH STUDY

**Site Principal Investigator:** Jie Li, PhD, RRT, RRT-ACCS, RRT-NPS

**Department:** Department of Cardiopulmonary Sciences, Division of

Respiratory Care

Address and Contact Information: 1620 W Harrison St, Tower LL1202, Chicago, IL. 60612.

Jie Li@rush.edu; 312-947-0065

**Protocol Title:** 

A Multicenter Randomized Controlled Trial of Early Use of Prone Positioning Combined with HFNC in COVID-19 Induced Moderate to severe Acute Respiratory Distress

Syndrome

Name of Participant:

RUSH

### **Key Information:**

IRB

You are being invited to participate in a research study. Research studies answer important questions that might help change or improve the way we do things in the future.

This consent form will give you information about the study to help you decide whether you want to participate. Please read this form, and ask any questions you have, before agreeing to be in the study.

Taking part in this research study is voluntary. You do not have to participate in this study and may choose to leave the study at any time. If you decide not to participate in this study or leave the study at a later time, your health care, benefits, or relationship with Rush University Medical Center will not change or be affected.

The purpose of this study is to investigate if early use of prone positioning combined with high-flow nasal cannula (HFNC) could improve oxygenation and ultimately avoid intubation in COVID-19 induced moderate to severe Acute Respiratory Distress Syndrome patients.

If you agree to participate in this study, your participation may last up to four weeks.

During these visits, you will be change your position to prone if you are randomized to prone position group.

There are risks to you for participating in this study. In this study, there is a risk of deterioration of hypoxia when you are turning to the prone position, but clinicians will monitor your saturation and titrate oxygen to meet your need to prevent hypoxemia. You may also have skin breakdown

Rush Template Version Date: 11/12/2019

Consent/Authorization Version Date: 03/31/2020 

during prone position, but your comfort will be checked by clinicians every 30 minutes, you are allowed to turn back to supine position any time you feel any discomfort.

You may benefit from taking part in this study. Based on experience with HFNC and prone positioning in patients with similar conditions, researchers believe it may be of benefit to people with your condition. However, because individuals respond differently to therapy, no one can know in advance if it will be helpful for you.

You have the option to not participate in this study.

Detailed Information: Please review the rest of this document for details about the above topics and additional information you should know before making a decision about whether or not you will participate in this study.

# Why are you being invited to participate in this study?

You are being asked to participate in this study because you are diagnosed as COVID-19 induced moderate to severe Acute Respiratory Distress Syndrome.

# How many participants will take part in this study?

Approximately 350 participants are expected to take part in this study. And 120 participants are expected to take part in the study at Rush.

# What are the activities you will be doing if you participate in this study?

If you agree to be in this study, you will be asked to participate in the following activities:

# **During the Screening Period**

You will receive high-flow nasal cannula oxygen therapy for 30 minutes to measure your oxygenation.

- During the Treatment Period
  You will be randomized to continue using high-flow nasal cannula oxygen therapy, or prone position with high-flow nasal cannula oxygen therapy.
  - If you assigned to the treatment of prone position with high-flow nasal cannula oxygen therapy, you will turn the position to prone by yourself at your pace, clinicians will stay bedside with you during the position change, oxygen flow will be adjusted based on your response to prone position. During prone position therapy, you still need to wear highflow nasal cannula oxygen therapy. You will turn from supine to prone position for at least 30 minutes twice a day.

#### What are the risks and discomforts of participating in this study?

Side effects, risks, and/or discomforts from participation in this study may include:

- In this study, there is a risk of deterioration of hypoxia when you are being turned to the prone position, but precautions will be taken to prevent this from happening.
- When you received high flow nasal cannula treatment, you may feel discomfort for the hot humidified oxygen flow, and we will adjust the temperature for you.

Rush Template Version Date: 11/12/2019

Consent/Authorization Version Date: 03/31/2020 

#### What if there is new information that may affect your decision to participate in this study?

During this study, you will be told about important findings (either good or bad), such as changes in the risks or benefits of participation in the study or new choices to participation that might cause you to change your mind about being in the study. If new information is shared with you, you may be asked to sign a revised consent form in order to continue participating in this study.

#### Will you receive your individual results from the study?

Generally, activities performed for research purposes are not meant to provide clinical information. We may learn things about you from this study which could be important to your health or treatment. If this happens, this information will be shared with you. You will know how your response to the treatment after you received the high-flow nasal cannula oxygen therapy or high-flow nasal cannula oxygen therapy plus prone positioning.

## Can you leave or be removed from this study?

You have the right to leave a study at any time without penalty. For your safety, however, you should consider the study doctor's advice about how to leave this study. If you leave this study before the final study visit, the study doctor may ask you to complete the final steps. You will receive the standard care if you decided to withdraw from the research.

The researchers and Sponsor also have the right to stop your participation in this study without your consent if:

- They believe it is in your best interests,
- You do not follow the instructions;
- The study is cancelled for any reason.

#### What about confidentiality of your medical information?

This authorization is voluntary. Rush University Medical Center and its affiliates ("Rush") will not withhold or refuse your treatment, payment, enrollment, or eligibility for benefits if you do not sign this authorization. You do not have to sign this authorization, but that means that you cannot be in the study or receive study-related treatment.

By signing this document, you voluntarily authorize (give permission to) Dr. Li, her study team, and other Rush personnel involved with the conduct and review of this study (which may include off-site personnel) to use or disclose (release) health information that identifies you for the study described in this document.

During the study, Dr. Li and her study team will collect Protected Health Information (PHI) about you for the purposes of this research. PHI is your health information that includes your medical history and new information obtained as a result of this study. Some of this information will come from your medical record. The health information that Rush may use or disclose for this research includes:

- Your demographic information, including age, gender, medical history, diagnosis for COVID-19;
- The laboratory and microbiology findings, treatment and outcome.

Rush Template Version Date: 11/12/2019

Consent/Authorization Version Date: 03/31/2020 

• Complications including skin breakdown, IV line or nasal cannula dislodgement or desaturation during position change.

• The respiratory assessments before, during the treatments of high-flow nasal cannula oxygen therapy or high-flow nasal cannula oxygen therapy plus prone positioning.

Dr. Li and her study team may share your health information and the results of your study-related procedures and tests with people outside of Rush who assist with the conduct and review of this study. The persons who receive your health information may not be required by Federal privacy laws to protect it and may share your information with others without your permission, but only if permitted by the laws governing them. Your health information described above may be used or disclosed to:

• Monitoring agencies such as the Food and Drug Administration (FDA), the National Institutes of Health and the Rush Institutional Review Board (IRB).

While you participate in the study you will have access to your medical record, but Dr. Li is not required to release to you study information that is not part of your medical record. Rush is required by law to protect your health information, and study records that identify you will be kept confidential. The results of study tests/procedures performed as part of this study may become part of your medical record. Any study information in your medical record will be kept indefinitely. Your identity will not be revealed on any report, publication, or at scientific meetings.

You have a right to inspect and copy the information to be disclosed with this authorization and you may obtain a copy of the information by contacting the office listed below.

If you no longer want to be in the study and do not want your future health information to be used, you may change your mind and revoke (take back) this authorization at any time by writing to Dr. Li at 1620 W Harrison St, Tower LL1202, Chicago, IL. 60612. If the authorization is revoked, you will no longer be allowed to participate in the study and previously authorized individuals/entities may still use or disclose health information that they have already obtained about you as necessary to maintain the integrity or reliability of the current study.

This authorization is valid for the entirety of this research study. It will expire upon completion of the study or if you revoke (take back) the authorization.

If you withdraw from this study, the data already collected from you may not be removed from the study records. The study doctor and/or study team may ask you whether they can continue to collect follow-up data on you. If follow-up information will be requested, you will be asked to sign a separate consent form before this information can be collected.

Records of participation in this study will be maintained and kept confidential as required by law. We will use coded names or identification numbers, removal of all identifying information.

The Rush Institutional Review Board (IRB) will have access to your files as they pertain to this research study. The IRB is a special committee that reviews new and ongoing human research

Rush Template Version Date: 11/12/2019

Consent/Authorization Version Date: 03/31/2020 

studies to check that the rules and regulations are followed regarding the protection of the rights and welfare of human participants.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. This research study can be found by searching for the following Clinical Trial Registry Number (NCT#): 04325906.

#### What are the costs to participate in this study?

There are no costs to you for participating in this research.

#### Will you be paid for your participation in this study?

You will not be paid for being in this study.

### SIGNATURE BY THE PARTICIPANT:

By signing below, you are consenting to participate in this research study. You have read the information given or someone has read it to you. You have had the opportunity to ask questions, which have been answered satisfactorily to you by the study staff. You do not waive any of your legal rights by signing this consent/authorization form. You will be given a signed copy of this document.

| 22 | IIVD | <b>■</b> £ |
|---|---|---|
| Name of Participant | Signature of Participan | Date of Signature |
| | Approved / | l j |
| Minor Assent | | Date of Signature |
| Parent, Guardian or Lega | al Representative's Signature | Date of Signature |
| SIGNATURE BY THE | INVESTIGATOR/INDIVIDUAL OBTA | INING CONSENT: |
| I attest that all the element | nts of informed consent described in this con | nsent document have been |
| • | chnical terms with the participant. I further a | attest that all questions asked |
| by the participant were a | nswered to the best of my knowledge. | |
| Signature of Individual Obtaining Consent | | Date of Signature |

Rush Template Version Date: 11/12/2019

Consent/Authorization Version Date: 03/31/2020 